CLINICAL TRIAL: NCT05333380
Title: Study on the Effectiveness of Atrial Fibrillation Analysis Software in Atrial Fibrillation Rhythm Monitoring
Brief Title: Study on the Effectiveness of AF Analysis Software in AF Rhythm Monitoring
Acronym: PPG-AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Heart Health Research Center (Other)
Responsible Party: Principal Investigator, Chang sheng Ma, Center Director, Beijing Anzhen Hospital
Other Study IDs: 2022-PPG-AF
Record Dates: First submitted 2022-04-01; First posted 2022-04-19 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation Paroxysmal
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ECG/PPG monitoring — The enrolled patients will wear an "ECG patch" and watch at the same time to collect ECG and PPG data respectively. The data collection time is from the day of hospitalization to before the ablation operation, and from 2 hours after the removal of ECG monitoring equipment to before leaving the hospital. The monitoring duration of each patient shall not be less than 18 hours.

SUMMARY:
Atrial fibrillation (AF) is a serious public health problem because of its increasing incidence and prevalence in the aging population. ECG is the most commonly used gold standard for clinical diagnosis of arrhythmias, but conventional ECG examinations are not adequate for long-term ECG follow-up measurements in patients with AF.

In this study, the AF patients will wear an watch and ECG patch to continuously monitor ECG and PPG. The software uses an integrated diagnostic mechanism of "AF burden + AF segments" to efficiently analyze ECG and PPG data, which can quickly and accurately identify the occurrence of AF and analyze AF burden in real-time, facilitating physicians' diagnosis and treatment and efficacy assessment.

DETAILED DESCRIPTION:
PPG-AF study is a Cohort randomized observational study.The trial will include patients with AF who meet the study requirements from Beijing Anzhen Hospital within 2 months. Each participant will wear an watch and ECG monitor after admission to hospital until Radiofrequency ablation for AF, and after AF ablation until discharge. And more than 18 hours in each period.

1. Primary endpoint. The ECG and PPG data are automatically analyzed by the AF analysis software. The results are compared with expert-annotated gold standard results to verify the sensitivity and specificity.
2. Secondary endpoints. The AF burden calculated from PPG data is compared with that from ECG monitoring, to verify the feasibility of daily monitoring of AF burden using PPG analysis.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age.
* Have clear ECG-recorded atrial fibrillation in the past and will undergo atrial fibrillation ablation in the current hospitalization.
* Patients who agree to wear both the watch and the ECG recorder.

Exclusion Criteria:

* Inability to wear the watch due to limited mobility or other problems.
* Severe skin diseases such as skin allergies or skin ulcers.
* Chronic insomnia not treated with medication.
* Patients with severe cardiovascular disease who may be resuscitated at any time.
* Previous history of Parkinson's, schizophrenia, epilepsy.
* Black people and those with excessively dark skin.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation who were hospitalized in the Department of Cardiology, Beijing Anzhen Hospital, aged from 18 to 80,were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 266 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
The ECG and PPG data are automatically analyzed by the AF analysis software. | Two months after enrollment of the first subject
  The results are compared with expert-annotated gold standard results to verify the sensitivity and specificity.

SECONDARY OUTCOMES:
The AF burden calculated from PPG data is compared with that from ECG monitoring. | Two months after enrollment of the first subject
  The AF burden calculated from PPG data is compared with that from ECG monitoring, to verify the feasibility of daily monitoring of AF burden using PPG analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374
- [Background] Wang Z, Chen Z, Wang X, Zhang L, Li S, Tian Y, Shao L, Hu H, Gao R; for China Hypertension Survey Group. The Disease Burden of Atrial Fibrillation in China from a National Cross-sectional Survey. Am J Cardiol. 2018 Sep 1;122(5):793-798. doi: 10.1016/j.amjcard.2018.05.015. Epub 2018 Jun 2. PMID 30049467
- [Background] Andrew NE, Thrift AG, Cadilhac DA. The prevalence, impact and economic implications of atrial fibrillation in stroke: what progress has been made? Neuroepidemiology. 2013;40(4):227-39. doi: 10.1159/000343667. Epub 2013 Jan 24. PMID 23364221
- [Background] Marini C, De Santis F, Sacco S, Russo T, Olivieri L, Totaro R, Carolei A. Contribution of atrial fibrillation to incidence and outcome of ischemic stroke: results from a population-based study. Stroke. 2005 Jun;36(6):1115-9. doi: 10.1161/01.STR.0000166053.83476.4a. Epub 2005 May 5. PMID 15879330
- [Background] Witassek F, Springer A, Adam L, Aeschbacher S, Beer JH, Blum S, Bonati LH, Conen D, Kobza R, Kuhne M, Moschovitis G, Osswald S, Rodondi N, Sticherling C, Szucs T, Schwenkglenks M; Swiss-AF study investigators. Health-related quality of life in patients with atrial fibrillation: The role of symptoms, comorbidities, and the type of atrial fibrillation. PLoS One. 2019 Dec 23;14(12):e0226730. doi: 10.1371/journal.pone.0226730. eCollection 2019. PMID 31869399
- [Background] McManus DD, Lee J, Maitas O, Esa N, Pidikiti R, Carlucci A, Harrington J, Mick E, Chon KH. A novel application for the detection of an irregular pulse using an iPhone 4S in patients with atrial fibrillation. Heart Rhythm. 2013 Mar;10(3):315-9. doi: 10.1016/j.hrthm.2012.12.001. Epub 2012 Dec 6. PMID 23220686
- [Background] Freedman B, Camm J, Calkins H, Healey JS, Rosenqvist M, Wang J, Albert CM, Anderson CS, Antoniou S, Benjamin EJ, Boriani G, Brachmann J, Brandes A, Chao TF, Conen D, Engdahl J, Fauchier L, Fitzmaurice DA, Friberg L, Gersh BJ, Gladstone DJ, Glotzer TV, Gwynne K, Hankey GJ, Harbison J, Hillis GS, Hills MT, Kamel H, Kirchhof P, Kowey PR, Krieger D, Lee VWY, Levin LA, Lip GYH, Lobban T, Lowres N, Mairesse GH, Martinez C, Neubeck L, Orchard J, Piccini JP, Poppe K, Potpara TS, Puererfellner H, Rienstra M, Sandhu RK, Schnabel RB, Siu CW, Steinhubl S, Svendsen JH, Svennberg E, Themistoclakis S, Tieleman RG, Turakhia MP, Tveit A, Uittenbogaart SB, Van Gelder IC, Verma A, Wachter R, Yan BP; AF-Screen Collaborators. Screening for Atrial Fibrillation: A Report of the AF-SCREEN International Collaboration. Circulation. 2017 May 9;135(19):1851-1867. doi: 10.1161/CIRCULATIONAHA.116.026693. PMID 28483832
- [Background] Perez MV, Mahaffey KW, Hedlin H, Rumsfeld JS, Garcia A, Ferris T, Balasubramanian V, Russo AM, Rajmane A, Cheung L, Hung G, Lee J, Kowey P, Talati N, Nag D, Gummidipundi SE, Beatty A, Hills MT, Desai S, Granger CB, Desai M, Turakhia MP; Apple Heart Study Investigators. Large-Scale Assessment of a Smartwatch to Identify Atrial Fibrillation. N Engl J Med. 2019 Nov 14;381(20):1909-1917. doi: 10.1056/NEJMoa1901183. PMID 31722151
- [Background] Wasserlauf J, You C, Patel R, Valys A, Albert D, Passman R. Smartwatch Performance for the Detection and Quantification of Atrial Fibrillation. Circ Arrhythm Electrophysiol. 2019 Jun;12(6):e006834. doi: 10.1161/CIRCEP.118.006834. PMID 31113234